CLINICAL TRIAL: NCT07291713
Title: Evaluating the Effects of an Online Positive Mental Health BMI Learning Program on Psychological Health in Patients With Myasthenia Gravis and Its Association With Adverse Childhood Experiences
Brief Title: Psychological Health and Adverse Childhood Experiences in Myasthenia Gravis: Online Mental Health BMI Learning Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jiann-Horng Yeh (Other)
Responsible Party: Sponsor-Investigator, Jiann-Horng Yeh, Vice Superintendent, Professor of Neurology, Shin Kong Wu Ho-Su Memorial Hospital, Shin Kong Wu Ho-Su Memorial Hospital
Organization: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20230731R
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Myasthenia Gravis; Adverse Childhood Experience; Psychological Well-being; Mental Well-being; Depressive Symptoms; Psychological Stress; Quality of Life (QOL); Activities of Daily Living; Emotional Regulation; Mental Health; Well-Being, Psychological
Keywords: myasthenia gravis; adverse childhood experience; online learning program; positive mental health BMI learning program; emotional regulation; emotional stability; psychological well-being; mental health BMI
MeSH Terms: conditions — Myasthenia Gravis; Psychological Well-Being; Depression; Stress, Psychological; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: All participants were enrolled into a single study group and received the same online behavioral intervention, the online Positive Mental Health BMI Learning Program. Pre-test and post-test assessments were completed by participants to measure psychological outcomes.
Masking Description: This was an open-label study in which no masking was used. All participants and investigators were aware of the behavioral intervention being provided.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): All participants were assigned to a single intervention arm and received the Positive Mental Health BMI Learning Program. This program consisted of four pre-recorded online video units delivered over four months through a closed Facebook group. The units covered interpersonal support, emotional regulation, and self-worth and meaning. Participants completed pre-test assessments before beginning the program and post-test assessments after completing all four units.
  Interventions: Behavioral: Positive Mental Health BMI Learning Program

INTERVENTIONS:
Behavioral: Positive Mental Health BMI Learning Program — The intervention consisted of the Positive Mental Health BMI Learning Program, a four-unit online behavioral program delivered through a closed Facebook group. Each video unit was approximately 15 minutes and focused on components of positive mental health, including interpersonal support, emotional regulation, and sense of meaning and self-worth. One unit was released each month over a four-month period. Participants completed pre-test assessments before the program and post-test assessments after completing all four units.

SUMMARY:
This study evaluated psychological health in patients with myasthenia gravis (MG) using an online behavioral program called the "Positive Mental Health BMI Learning Program." The program consisted of four short video units focused on interpersonal support, emotional regulation, and personal meaning. Patients receiving care in the neurology outpatient clinic were invited to complete questionnaires before and after viewing the online program. Psychological well-being, depressive symptoms, daily functioning, and quality of life were assessed to describe participants' mental health status and changes observed over the course of the program.

DETAILED DESCRIPTION:
Participants completed sociodemographic questionnaires, adverse childhood experiences (ACEs) assessments, and four psychological and disease-related measures: the Myasthenia Gravis Activities of Daily Living Scale (MG-ADL), the Myasthenia Gravis Quality of Life 15-item scale (MG-QOL15), the mental health BMI indicator (mBMI), and the Patient Health Questionnaire-9 (PHQ-9). The study collected baseline data prior to the online program and post-intervention data after completion of the four video units. Analyses examined associations between ACE exposure and psychological measures, as well as changes in clinical and psychological indicators across the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of myasthenia gravis (MG) based on acetylcholine receptor antibody testing, single-fiber electromyography, repetitive nerve stimulation, or chest computed tomography.
* Individuals able to clearly express their own intentions.
* Individuals without cognitive impairment or psychiatric disorders.
* Individuals who are able to use Facebook and who agree to participate in the study and provide written informed consent.

Exclusion Criteria:

* Individuals who do not have a diagnosis of MG.
* Patients who are unable to communicate adequately in Mandarin, Taiwanese, English, or written form.
* Individuals with head trauma, psychiatric symptoms, or cognitive impairment that may interfere with verbal expression.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2025-01-09 (Actual); Study Completion 2025-01-09 (Actual)

PRIMARY OUTCOMES:
Change in the indicator of mental health BMI on well-being (mBMI) Score from baseline to post-intervention | Baseline to 4 months
  The indicator of mental health BMI (mBMI) is a measure of positive psychological well-being that includes three domains:
  1. Befriend (B), representing interpersonal support and closeness
  2. Mindfulness (M), representing emotional stability and awareness
  3. Identity (I), representing self-worth and meaning.
  Scores were collected before the intervention and after completion of the four-unit online program to evaluate changes in psychological well-being.

SECONDARY OUTCOMES:
Change in Patient Health Questionnaire-9 (PHQ-9) Score from baseline to post-intervention | Baseline to 4 months
  The Patient Health Questionnaire-9 (PHQ-9) is a 9-item measure used to assess the severity of depressive symptoms. Participants completed the PHQ-9 before the intervention and again after completing the four-unit online program to evaluate changes in depressive symptom severity over time.
Change in Myasthenia Gravis Quality of Life 15-item (MG-QOL15) Score from baseline to post-intervention | Baseline to 4 months
  The Myasthenia Gravis Quality of Life 15-item scale (MG-QOL15) is a disease-specific measure used to assess the impact of myasthenia gravis on daily functioning and overall quality of life. Participants completed the MG-QOL15 before the intervention and again after completing the four-unit online program to evaluate changes in disease-related quality of life.
Change in Myasthenia Gravis Activities of Daily Living (MG-ADL) Score from baseline to post-intervention | Baseline to 4 months
  The Myasthenia Gravis Activities of Daily Living scale (MG-ADL) is an 8-item measure used to assess symptom severity and the impact of myasthenia gravis on daily functioning. Participants completed the MG-ADL before the intervention and again after completing the four-unit online program to evaluate changes in disease-related functional status.

CONTACTS AND LOCATIONS:
Overall Officials: Jiann-Horng Yeh, MD, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data.

REFERENCES:
- [Background] Liu, S. M. (2020). The Study of Cut-off Scores for Mental Health BMI Index. [master's thesis]. [Taipei (Taiwan, R.O.C.)]: National Taipei University of Nursing and Health Sciences. Available at: https://hdl.handle.net/11296/p992dy
- [Background] Li, Y. C. (2019). The Cluster Analysis of the Positive and Negative Indicators of Complete Mental Health State Model. Special Research of the Ministry of Science and Technology (MOST 108-2637-H-227-001). Available at: https://www.airitilibrary.com/Article/Detail?DocID=U0068-0309202111314000
- [Background] Li, Y. C. and Chen, Y. F. (2016). National mental health BMI. Couns. Guid. 369, 50-55. doi: 10.6251/bep.202406_55(4).0008
- [Background] Li, Y. C., Fang, C. K., Liu, C. Y., and Chang, W. H. (2024). Cluster Analysis of the Positive and Negative Indicators of Complete Mental Health State Model. Chinese Journal of Guidance and Counseling, 69, 37-75. Chin. J. Guid. Couns. 69, 37-75. doi: 10.53106/172851862024010069002
- [Background] Harris, N. B. (2018). The Deepest Well: Healing the Long-Term Effects of Childhood Adversity. New York, NY: Houghton Mifflin Harcourt. ISBN-13: 978-0544828704
- [Background] Chiu, T. Y. (2021). Effect of Promoting Positive Mental Health BMI by Group Counseling for Myasthenia Gravis. [master's thesis]. [Taipei (Taiwan, R.O.C.)]: National Taipei University of Nursing and Health Sciences. Available at: https://hdl.handle.net/11296/62vwcp
- [Background] Chung, M. Y. (2018). Building Mental Health BMI Indicator on Well-Being: A Sampling from Myasthenia Gravis Patients. [master's thesis]. [Taipei (Taiwan, R.O.C.)]: National Taipei University of Nursing and Health Sciences. Available at: https://hdl.handle.net/11296/st3u9u
- [Background] Chen, Y. J. (2023). The relationships among adverse childhood experiences, resilience, and health status in patients with ankylosing spondylitis. [master's thesis]. [Taichung (Taiwan, R.O.C.)]: Chung Shan Medical University. Available at: https://hdl.handle.net/11296/d55q94
- [Background] Liao, C. M. (2022). A Relational Research on Personality Traits, Resilience, and Career Self-Efficacy among Adults with Adverse Childhood Experiences. [master's thesis]. [Taipei (Taiwan, R.O.C.)]: National Taiwan Normal University. Available at: https://hdl.handle.net/11296/p3359x
- [Background] Huang, C. C. (2017). A Study on the Childhood Adversity Experiences and Resilience. [master's thesis]. [Kaohsiung (Taiwan, R.O.C.)]: Shu-Te University. Available at: https://hdl.handle.net/11296/d383p6
- [Background] Bellis MA, Hughes K, Ford K, Butler N, Wilson C, Quigg Z. Relative and combined contributions of adverse childhood experiences and self-reported child poverty to health and economic outcomes in adults - a retrospective study in a UK region. BMC Public Health. 2025 Oct 15;25(1):3501. doi: 10.1186/s12889-025-23938-z. PMID 41094458
- [Background] Bunting L, Davidson G, McCartan C, Hanratty J, Bywaters P, Mason W, Steils N. The association between child maltreatment and adult poverty - A systematic review of longitudinal research. Child Abuse Negl. 2018 Mar;77:121-133. doi: 10.1016/j.chiabu.2017.12.022. Epub 2018 Jan 12. PMID 29346067
- [Background] Liu SI, Yeh ZT, Huang HC, Sun FJ, Tjung JJ, Hwang LC, Shih YH, Yeh AW. Validation of Patient Health Questionnaire for depression screening among primary care patients in Taiwan. Compr Psychiatry. 2011 Jan-Feb;52(1):96-101. doi: 10.1016/j.comppsych.2010.04.013. Epub 2010 Jul 1. PMID 21111406
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Burns TM, Conaway MR, Cutter GR, Sanders DB; Muscle Study Group. Less is more, or almost as much: a 15-item quality-of-life instrument for myasthenia gravis. Muscle Nerve. 2008 Aug;38(2):957-63. doi: 10.1002/mus.21053. PMID 18642357
- [Background] Mullins LL, Carpentier MY, Paul RH, Sanders DB; Muscle Study Group. Disease-specific measure of quality of life for myasthenia gravis. Muscle Nerve. 2008 Aug;38(2):947-56. doi: 10.1002/mus.21016. PMID 18697209
- [Background] Wolfe GI, Herbelin L, Nations SP, Foster B, Bryan WW, Barohn RJ. Myasthenia gravis activities of daily living profile. Neurology. 1999 Apr 22;52(7):1487-9. doi: 10.1212/wnl.52.7.1487. PMID 10227640
- [Background] Felitti VJ, Anda RF, Nordenberg D, Williamson DF, Spitz AM, Edwards V, Koss MP, Marks JS. Relationship of childhood abuse and household dysfunction to many of the leading causes of death in adults. The Adverse Childhood Experiences (ACE) Study. Am J Prev Med. 1998 May;14(4):245-58. doi: 10.1016/s0749-3797(98)00017-8. PMID 9635069